CLINICAL TRIAL: NCT06857201
Title: Randomized Assessment of Left Bundle Branch Area Pacing Versus Right Ventricular Pacing in Post-TAVR Patients with Persistent High-Degree Atrioventricular Block or Complete Heart Block Requiring Permanent Pacemaker Implantation
Brief Title: RAFT-TAVR PACE: LBBAP Vs. RVP Post-TAVR in Patients Requiring PPI
Acronym: RAFT-TAVR PACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Habib Khan, Dr. Habib Khan, Co-Principal Investigator, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5143
Record Dates: First submitted 2025-02-06; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-12

CONDITIONS: High Degree Second Degree Atrioventricular Block; Complete Heart Block; Heart Failure; Transcatheter Aortic Valve Replacement (TAVR); Conduction Disorder
Keywords: Left Bundle Branch Area Pacing (LBBAP); Right Ventricular Pacing (RVP); Transcatheter Aortic Valve Replacement (TAVR); Permanent Pacemaker Implantation (PPI); High-Degree Atrioventricular Block (HDAVB); Complete Heart Block (CHB); Conduction System Pacing (CSP); Heart Failure; cardiovascular mortality; Ventricular Dyssynchrony; Pacing-Induced Cardiomyopathy; Electrophysiology; cardiac pacing; Physiological Pacing; ventricular function; Left Ventricular Ejection Fraction (LVEF); Clinical Outcomes Post-TAVR; Quality of Life (QoL); Aortic Stenosis; Heart Rhythm Disorders
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac; Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Left Bundle Branch Area Pacing (LBBAP) Group (Experimental): Participants randomized to receive Left Bundle Branch Area Pacing (LBBAP) after Transcatheter Aortic Valve Replacement (TAVR). This pacing technique aims to preserve physiologic ventricular activation by directly pacing the left bundle branch area.
  Interventions: Procedure: Left Bundle Branch Area Pacing
- Right Ventricular Pacing (RVP) Group (Active Comparator): Participants randomized to receive Right Ventricular Pacing (RVP) after Transcatheter Aortic Valve Replacement (TAVR). This technique is the traditional pacing method, which stimulates the right ventricle to maintain cardiac rhythm.
  Interventions: Procedure: Right Ventricular Pacing

INTERVENTIONS:
Procedure: Left Bundle Branch Area Pacing — LBBAP is performed during permanent pacemaker implantation post-TAVR.
  Arms: Left Bundle Branch Area Pacing (LBBAP) Group
Procedure: Right Ventricular Pacing — RVP is performed during permanent pacemaker implantation post-TAVR.
  Arms: Right Ventricular Pacing (RVP) Group

SUMMARY:
The RAFT-TAVR PACE study is a clinical trial designed to compare two types of heart pacing methods in patients who develop conduction problems after undergoing a transcatheter aortic valve replacement (TAVR) procedure.

This study will evaluate whether Left Bundle Branch Area Pacing (LBBAP), a newer and more natural pacing method, is better than the traditional Right Ventricular Pacing (RVP) at improving heart function and patient outcomes.

The study aims to recruit 60 patients across six centers and will focus on the safety, feasibility, and success of LBBAP compared to RVP. Patients will be followed for one year to assess heart function, quality of life, and any complications related to the pacing method.

DETAILED DESCRIPTION:
The RAFT-TAVR PACE study is a multi-center, double-blind, randomized controlled trial (RCT) designed to compare Left Bundle Branch Area Pacing (LBBAP) and Right Ventricular Pacing (RVP) in patients who develop persistent high-degree atrioventricular block (HDAVB) or complete heart block (CHB) following Transcatheter Aortic Valve Replacement (TAVR).

Background & Rationale:

TAVR is an established treatment for severe aortic stenosis, but conduction disturbances requiring permanent pacemaker implantation (PPI) remain a common complication, affecting approximately 15-25% of patients post-TAVR. Conventional RVP has been associated with ventricular dyssynchrony, adverse cardiac remodeling, and increased risk of heart failure.

LBBAP is an emerging conduction system pacing technique that may preserve physiological ventricular activation by engaging the His-Purkinje system more effectively. While observational studies suggest LBBAP may improve ventricular function, quality of life, and clinical outcomes compared to RVP, no large-scale RCT has yet validated these benefits in post-TAVR patients requiring PPI.

Study Objectives:

Primary Objective: Assess the feasibility and success rate of LBBAP implantation in post-TAVR patients requiring PPI and determine if LBBAP results in improved outcomes over RVP.

Secondary Objectives: Evaluate the impact of LBBAP versus RVP on:

Left ventricular activation Left ventricular ejection fraction (LVEF) Quality of life (KCCQ, EQ-5D-5L) Heart failure events and adverse clinical outcomes

Study Design:

The Vanguard Phase will enroll 60 patients across six sites over nine months to establish the feasibility, procedural success, and safety of LBBAP. If successful, the study will expand into a full-scale RCT.

Randomization (1:1) occurs after the clinical decision to implant a pacemaker post-TAVR.

Blinding: The study is double-blinded-patients and follow-up clinicians are blinded to pacing allocation. The implanting physician is unblinded for procedural purposes.

Follow-up Duration: 12 months, with scheduled assessments at 3, 6, and 12 months, including pacemaker interrogation, echocardiography, and quality-of-life questionnaires.

Key Endpoints:

Primary Endpoint:

Feasibility of recruitment (60 patients in 9 months) LBBAP implantation success rate >90%

Secondary Endpoints:

Improvement in left ventricular activation LVEF at 12 months Quality of life (KCCQ, EQ-5D-5L) changes Rates of heart failure hospitalization and adverse events

Safety & Data Monitoring:

An independent Data and Safety Monitoring Board (DSMB) will oversee patient safety.

Adverse events will be adjudicated by a blinded committee and reported per regulatory guidelines.

Data collection will be managed through a secure REDCap database.

Significance:

This study will generate critical evidence to determine whether LBBAP should be the preferred pacing modality for post-TAVR patients requiring PPI. If proven superior, LBBAP could redefine post-TAVR pacing guidelines, improving patient outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Successful insertion of TAVR for aortic stenosis
2. Persistent HDAVB or CHB identified within 30 days of TAVR

   ● HDAVB is defined as any of the following(9): Second-degree AV block type 2 (Mobitz II) in the presence of a QRS ≥120 msec, or 2:1 AV block in the presence of a QRS ≥120 msec, or ≥2 consecutive P waves at a constant physiologic rate that do not conduct to the ventricles, or transient third-degree AV block, or in the setting of AF a prolonged pause (>3 s) or a fixed slow (<50 beats/min) ventricular response rate.
3. Age ≥ 18 years

Exclusion Criteria:

1. Patients with a pacemaker/ICD/CRT prior to TAVR
2. More than mild para-valvular regurgitation following TAVR
3. Patients with clinical indication for CRT-D or CRT-P
4. Patients with mechanical tricuspid valve
5. Renal failure - eGFR<15 or on dialysis
6. Un-revascularized coronary artery disease with proximal multi-vascular coronary disease
7. Acute coronary syndrome with 3 months
8. Cardiogenic shock requiring inotropic therapy within 1 week
9. Life-expectancy < 2 years
10. Anticipating heart transplant within 1 year
11. Pregnant or intending to become pregnant within the study period
12. Participating in another randomized controlled trial
13. Unable or unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-09-26 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
CV Mortality and Heart Failure Events | from enrollment to the 12 month FU at minimum, with data collected every 6 months after until study completion at 5 year mark
  The primary outcome of the full-scale RCT is a composite of CV mortality and HF events. All deaths and in-patient/outpatient unscheduled encounters will be adjudicated by a clinical events adjudication committee. HF events are defined as an admission to a healthcare facility for >24 hours with a diagnosis of worsening HF or worsening HF requiring intravenous HF therapy and ultrafiltration at an urgent or outpatient healthcare facility.
  The rationale for using CV mortality and HF events as the primary outcome is that pacing therapy will not prevent non-CV deaths. The rationale for including the worsening of HF managed in outpatient facilities is that more patients are managed aggressively with IV diuretics in emergency departments, HF clinics, and infusion centers, avoiding hospitalization. This is accepted by Health Canada, US Food and Drug Administration, and European Medicines Agency.
Successful Enrollment and Randomization | from start of enrollment to end of vanguard/pilot phase of study, enrolling 60 patients
  (1) Successfully enroll and randomize 60 patients in 9 months from 6 participating centers
VANGUARD - Successful implantation of devices | Vanguard phase - from enrollment to the 60th patient being enrolled and followed up at 12 month FU point
  (2) Successfully implant the devices in 60 randomized patients, defined as <10% inability to implant LBBAP lead in those randomized to have LBBAP
VANGUARD - at least 90% ventricular pace at 3 months follow up | enrollment to 3 month FU timepoint
  >90% ventricular pace in these 60 patients at 3 months follow-up

SECONDARY OUTCOMES:
CV Mortality | at least 12 months until 4 years when the study is complete and all data is collected for the last participant
  Compare the incidence of cardiovascular mortality between the LBBAP and RVP groups over the entire follow-up period of the study.
Heart Failure Events | minimum 1 year to end of study completion, average of 5 years
  Compare the incidence of heart failure events, including heart failure hospitalizations, between the LBBAP and RVP groups during the entire follow-up period.
Quality of Life Assessment Change | enrollment to end of study completion, an average of 5 years
  Change of Quality-of-Life assessment Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline
Change of NT-proBNP | 1 year
  Change of NT-proBNP from baseline
Left Ventricular Ejection Fraction (LVEF) | 1 year
  Measure and compare changes in LVEF between LBBAP and RVP groups using echocardiographic assessments.
Quality of Life Assessment Change - EQ5D | from baseline enrollment to end of study, average of 5 years
  Change of Quality-of-Life assessment EQ5D from baseline

OTHER OUTCOMES:
Device-related hospitalization | 1 year
  Assess the incidence of hospitalizations directly related to the implanted device in both the LBBAP and RVP groups.
Device Implant-Related Complications | 1 year
  Evaluate the occurrence of device-related complications requiring medical or surgical intervention, including:
  1. Pocket infection requiring hospitalization or surgical intervention.
  2. Lead dislodgement requiring repositioning or replacement.
  3. Cardiac tamponade requiring intervention.
  4. Device pocket issues, including hematoma requiring intervention.

IPD SHARING:
Plan to Share IPD: Undecided